CLINICAL TRIAL: NCT04178070
Title: A Randomized, Double-blind, Placebo-controlled, Single Dose, Dose-escalated Phase Ⅰ Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Gerilimzumab in Healthy Adult Subjects.
Brief Title: Phase Ⅰ Clinical Trial of Gerilimzumab Injection in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GENOR GB224-001; V1.4
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- GB224 2mg (Experimental): single dose
  Interventions: Biological: GB224 2mg
- GB224 5mg (Experimental): single dose
  Interventions: Biological: GB224 5mg
- GB224 10mg (Experimental): single dose
  Interventions: Biological: GB224 10mg
- GB224 15mg (Experimental): single dose
  Interventions: Biological: GB224 15mg
- GB224 20mg (Experimental): single dose
  Interventions: Biological: GB224 20mg
- GB224 30mg (Experimental): single dose
  Interventions: Biological: GB224 30mg; Other: Placebo, 30mg
- Placebo 2mg (Placebo Comparator): single dose
  Interventions: Other: Placebo, 2mg
- Placebo 5mg (Placebo Comparator): single dose
  Interventions: Other: Placebo, 5mg
- Placebo 10mg (Placebo Comparator): single dose
  Interventions: Other: Placebo, 10mg
- Placebo 15mg (Placebo Comparator): single dose
  Interventions: Other: Placebo, 15mg
- Placebo 20mg (Placebo Comparator): single dose
  Interventions: Other: Placebo, 20mg
- Placebo 30mg (Placebo Comparator): single dose
  Interventions: Other: Placebo, 30mg

INTERVENTIONS:
Biological: GB224 2mg — 2mg (100μL), single dose, abdominal subcutaneous injection
  Other Names: Gerilimzumab injection
  Arms: GB224 2mg
Biological: GB224 5mg — 5mg (250μL), single dose, abdominal subcutaneous injection
  Other Names: Gerilimzumab injection
  Arms: GB224 5mg
Biological: GB224 10mg — 10mg (500μL), single dose, abdominal subcutaneous injection
  Other Names: Gerilimzumab injection
  Arms: GB224 10mg
Biological: GB224 15mg — 15mg (750μL), single dose, abdominal subcutaneous injection
  Other Names: Gerilimzumab injection
  Arms: GB224 15mg
Biological: GB224 20mg — 20mg (1mL), single dose, abdominal subcutaneous injection
  Other Names: Gerilimzumab injection
  Arms: GB224 20mg
Biological: GB224 30mg — 30mg (1.5mL), single dose, abdominal subcutaneous injection
  Other Names: Gerilimzumab injection
  Arms: GB224 30mg
Other: Placebo, 2mg — 2mg (100μL), single dose, abdominal subcutaneous injection
  Arms: Placebo 2mg
Other: Placebo, 5mg — 5mg (250μL), single dose, abdominal subcutaneous injection
  Arms: Placebo 5mg
Other: Placebo, 10mg — 10mg (500μL), single dose, abdominal subcutaneous injection
  Arms: Placebo 10mg
Other: Placebo, 15mg — 15mg (750μL), single dose, abdominal subcutaneous injection
  Arms: Placebo 15mg
Other: Placebo, 20mg — 20mg (1mL), single dose, abdominal subcutaneous injection
  Arms: Placebo 20mg
Other: Placebo, 30mg — 30mg (1.5mL), single dose, abdominal subcutaneous injection
  Arms: GB224 30mg; Placebo 30mg

SUMMARY:
The primary objectives of this study are to evaluate the safety, tolerability and pharmacokinetic (PK) profiles of single-dose, dose-escalated, abdominal subcutaneous injection of GB224 in Chinese healthy adult subjects. The secondary objectives are to preliminarily understand the immunogenicity and pharmacodynamic variable (IL-6) of single abdominal subcutaneous injection of GB224 in Chinese healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study procedures and contents, and voluntarily sign the informed consent form;
2. Chinese healthy adult volunteers aged 18 to 45 years, males and females;
3. The subjects have qualified physical examination within 30 days before the study, the body mass index (BMI) is within the range of 19~24 and the body weight is within the range of 45~75kg;
4. Males or females agree to adopt medically confirmed effective contraceptive measures during the entire study period and within 6 months after the end of this study.
5. The investigator considers that the patients have good health condition according to the physical examination, medical history, vital signs and ECG etc.
6. Patients have good compliance, can receive follow-up visits as scheduled, are able to well communicate with the investigators and complete the study as required by the study.

Exclusion Criteria:

1. Any of the following is met: allergic constitution; known allergic to the components of the investigational product or allergy history to any drug or food or pollen; subjects who have medical history of skin allergy such as physical urticaria; subjects who have abnormal serum immunoglobulin E (IgE) test;
2. Any of the current symptoms, signs or laboratory test abnormalities indicating the possible presence of acute or subacute infection (e.g., pyrexia, cough, urgent micturition, urodynia, abdominal pain, diarrhea, cutaneous infected wound etc.)
3. Patients with active pulmonary tuberculosis; patients who previously had medical history of active pulmonary tuberculosis;
4. Subjects who have medical history of drug addiction or drug abuse;
5. Subjects who have clear medical history of central nervous system, cardiovascular, renal, hepatic, gastrointestinal, respiratory, metabolic system or subjects with other significant diseases; subjects with medical history of hypertension or screening systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg, which are clinically significant at the discretion of the investigators; subjects who have medical history of orthostatic hypotension;
6. Subjects who have medical history of malignant tumors;
7. Subjects who participated in other clinical studies within 3 months before enrollment, or subjects who received drugs which are known to injure the major organs within 3 months before enrollment;
8. Subjects who used prescription drugs or non-prescription drugs within 14 days before enrollment;
9. Subjects who have blood donation history within 3 months before enrollment;
10. Subjects who meet any of the following criteria: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5 times the upper limit of normal (ULN), serum creatinine (Cr) > the upper limit of normal (ULN);
11. Abnormal routine blood tests: any of the following is met: white blood cells (WBC)<3.0×109/L or >9.5×109/L, neutrophil count (ANC)<1.5×109/L, platelet count (PLT)<100×109/L, hemoglobin (HGB)<104g/L;
12. Any of the following is positive: hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), acquired immunodeficiency syndrome antibody (Anti-HIV) and anti-treponema pallidum antibody (TP-Ab);
13. Subjects who have positive tuberculosis skin test (5 units of dosage, induration of not less than 5 millimeters (mm) within 48 ~ 72 hours);
14. Subjects with positive anti-nuclear antibody (ANA), anti-double stranded DNA antibody (ds-DNA) and anti-extractable nuclear antigens (ENA);
15. Subjects with positive anti-drug antibody (ADA);
16. Subjects with positive tumor markers (CEA, AFP, PSA and CA-125);
17. Subjects with abnormal coagulation function, which is clinically significant at the discretion of the investigators;
18. Subjects with medical history of psychiatric disorders;
19. Smoking more than 5 cigarettes/day or equivalent tobacco;
20. Weekly alcohol consumption more than 28 units (1 unit = 285 mL of beer or 25 mL of spirits or a glass of wine); or subjects who have positive breath alcohol test within 24 hours before the use of investigational drug;
21. Subjects who have clinically significant abnormal laboratory test values at screening;
22. Female subjects who have positive serum/urine pregnancy tests at screening or lactating women;
23. Patients who have insufficient communication, understanding and cooperation; or patients who have poor compliance and cannot guarantee to strictly follow the study protocol;
24. Subjects who are considered unsuitable for participating in this study for various reasons at the discretion of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Adeverse Effect, AE | Up to 112 days.
  Adeverse Effect, AE
Serious Adeverse Effect, AE | Up to 112 days.
  Serious Adeverse Effect, AE
Maximum Tolerated Dose, MTD | Up to 112 days.
  Maximum Tolerated Dose, MTD
Dose Limited Toxicity, DLT | Up to 112 days.
  Dose Limited Toxicity, DLT

SECONDARY OUTCOMES:
AUC0-t | Up to 112 days.
  AUC0-t
Cmax | Up to 112 days.
  Cmax
AUC0-∞ | Up to 112 days.
  AUC0-∞
Tmax | Up to 112 days.
  Tmax
Vd | Up to 112 days.
  Vd
Ke | Up to 112 days.
  Ke
Mean Retention Time, MRT | Up to 112 days.
  Mean Retention Time, MRT
t1/2 | Up to 112 days.
  t1/2
CL | Up to 112 days.
  CL

CONTACTS AND LOCATIONS:
Overall Officials: Yi Fang, Ph.D, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China